CLINICAL TRIAL: NCT00369239
Title: Is Premorbid Functioning a Predictor of Outcome in Patients With Early Onset Psychosis Treated With Risperdal Consta?
Brief Title: Treatment With Risperidone Long Acting Injectable (RLAI) in an Early Phase of Psychosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002263
Record Dates: First submitted 2006-08-25; First posted 2006-08-29 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia; Psychotic Disorders; Schizoaffective Disorder
Keywords: Early psychosis; premorbid functioning; Scale for Assessment of Insight; Risperdal Consta; risperidone long acting injectable
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

INTERVENTIONS:
Drug: risperidone long acting injectable

SUMMARY:
The purpose of this research study is to see how well patients in an early phase of their illness respond to treatment and whether this depends on how well they functioned socially, academically and vocationally before becoming ill. The study also examines whether patients with more insight into their illness have better outcomes.

DETAILED DESCRIPTION:
Intervention with antipsychotic medications during the early stages of schizophrenia may result in a better outcome for patients, with a higher number of patients achieving full remission, a shorter time to remission and decreased risk of relapse. In addition, there is evidence to suggest that a critical window of opportunity exists in the early period of syndromal differentiation, when pharmacological intervention and intensive engagement of the patient may impact favourably on symptoms in the longer term.

The long-acting injectable formulation of risperidone has shown improvements in measures of disease severity over the oral formulation, and demonstrated an improved safety and tolerability profile because of its lower peak-trough levels. A recent study has demonstrated that patients in the early phase of their illness (0-3 years) benefit from treatment with RLAI.

Although premorbid functioning is accepted to be a predictor of outcome and to affect treatment adherence, prospective clinical data are scarce. RLAI addresses the problem of adherence by eliminating the need for daily medication intake. In this study we investigate whether patients with good premorbid functioning respond better to treatment with RLAI compared to patients with poor premorbid functioning. Moreover, patients with schizophrenia often fail to acknowledge their illness and need for treatment - so-called 'lack of insight'. Previous studies investigating the relationship between acute psychopathology and insight have produced conflicting results. Multiple administrations of a structured measure of insight (SAI-E) and symptom measures will provide here a means to evaluate whether insight is correlated with clinical change, whether insight changes over time and whether changes in insight are related to changes in psychopathology.

A physical examination will be performed, including heart rate, blood pressure, and weight. Interviews and assessments will be made to complete standard rating scales (Positive and Negative Symptom Score (PANSS), Scale for Assessment of Insight-Expanded version (SAI-E), Clinical Global Impression (CGI), Global Assessment of Functioning (GAF), and Extrapyramidal Symptom Rating Scale (ESRS)). The Short-Form-36 questionnaire (SF-36) will be completed by the patient. Any health problems and medicines of the patient will be recorded.

The primary hypothesis, that patients with "Stable-good" premorbid functioning will have better outcomes than those with "Stable-poor" premorbid functioning will be examined by dividing patients into a "Stable-good" and "Stable-poor" premorbid functioning groups based on their total scores on the Premorbid Adjustment Scale (PAS). Statistically significant differences between the "Stable-good" vs. "Stable-poor" pre-morbid groups on the combined change measure at the 5% level will be interpreted as supporting the hypothesis.

Association of insight and outcomes will be examined using Scale for Assessment of Insight-Expanded version (SAI-E )and insight item (G 12) from Positive and Negative Symptom Score (PANSS). Effectiveness [Clinical Global Impression (CGI-S/C), PANSS, retention rate), functioning [Short-Form-36 questionnaire (SF-36, rehospitalisation rates)] and safety and tolerability will be assessed. The observation period is 6 months. RLAI is given as intramuscular injections every 2 weeks. The starting dose of RLAI will be in accordance with the product label (usually 25 mg). If necessary, the dosage of the injection may be increased gradually. Treatment duration is 26 weeks. To ensure continued antipsychotic coverage until the main release of risperidone from the microspheres, previous antipsychotic therapy will be continued concomitantly during the first three weeks of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia/schizoaffective disorder for no longer than 2 years
* At least 2 previous psychotic episodes
* At least 6 months of antipsychotic treatment required
* maximum total Positive and Negative Symptom Score (PANSS) score of < = 80
* Patients may be currently treated with any antipsychotic (with the exception of clozapine and depot neuroleptics) at doses not exceeding the registered highest recommended dose.

Exclusion Criteria:

* Already on treatment with RLAI
* Patients requiring treatment at entry with mood stabilizers or antidepressants may enter the study only if a stable dose has been received for 3 months prior to study entry
* Previously received treatment with clozapine
* Known non-responders to previous treatment with at least 2 antipsychotics
* Mental retardation
* Patients with conditions and symptoms that are listed in the SmPC under special warnings and special precautions for use
* Acute risk of suicide in the investigator's opinion at study entry or history of suicidal attempt(s) in the last 3 months before the study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2006-03; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To assess the use of RLAI in patients in the early phases of psychosis and to test the hypothesis that patients with good vs. poor premorbid functioning will have better treatment response over 6 months as assessed with the Premorbid Adjustment Scale.

SECONDARY OUTCOMES:
The association of insight and outcomes will be examined using SAI-E and insight item (G 12) from PANSS. Effectiveness (CGI-S/C, PANSS, retention rate), functioning (SF-36, rehospitalisation rates) and safety and tolerability will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.

REFERENCES:
- See also: Risperdal� Consta�: Clinical Study Report Synopsis RIS-SCH-4043 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=376&filename=CR002263_CSR.pdf